CLINICAL TRIAL: NCT03131050
Title: A Double-blind, Controlled, Randomized Study Comparing Escitalopram Combined With Scopolamine or Escitalopram in Patients With Major Depressive Disorder
Brief Title: Effectiveness Study of Scopolamine Combined With Escitalopram in Patients With MDD
Acronym: SCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Gang Wang, MD, Director of Beijing Anding Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Scopolamine i.m.
Record Dates: First submitted 2017-04-18; First posted 2017-04-27 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Major Depressive Disorder
Keywords: Scopolamine
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Scopolamine; Escitalopram; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: GROUP 1: The patients received intramuscular injection treatment of scopolamine (0.3 mg/ml) at 9 am and 0.9% saline treatment at 3pm. GROUP 2: The patients received intramuscular injection treatment of scopolamine (0.3 mg/ml) at 9 am and 3 PM. GROUP 3: The patients received intramuscular injection treatment of 0.9% saline (1 ml) at 9 am and 3 PM.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High-dose scopolamine add-on therapy (Experimental): Scopolamine (0.3 mg/1 ml, i.m.) Bid; escitalopram （10 mg/d p.o.）QD
  Interventions: Drug: Scopolamine; Drug: Escitalopram
- Low-dose scopolamine add-on therapy (Experimental): Scopolamine (0.3 mg/1 ml, i.m.) QD; placebo (1 ml saline, i.m.) QD; escitalopram （10 mg/d p.o.）QD
  Interventions: Drug: Scopolamine; Drug: Escitalopram; Drug: Saline
- Placebo add-on therapy (Placebo Comparator): Placebo (1 ml saline, i.m.) Bid; escitalopram （10 mg/d p.o.）QD
  Interventions: Drug: Escitalopram; Drug: Saline

INTERVENTIONS:
Drug: Scopolamine — Intramuscular injection with scopolamine (0.3 mg/1ml,QD or Bid) during the first three days;
  Arms: High-dose scopolamine add-on therapy; Low-dose scopolamine add-on therapy
Drug: Escitalopram — Oral escitalopram 10 mg/d throughout the total of 4 weeks treatment
Drug: Saline — Intramuscular injection with saline (1ml, QD or Bid) during the first three days;
  Arms: Low-dose scopolamine add-on therapy; Placebo add-on therapy

SUMMARY:
Despite the availability of a wide range of antidepressant drugs, clinical trials indicate that 30% to 40% of patients with major depression fail to respond to first-line antidepressant treatment, despite adequate dosage, duration, and compliance. Moreover, in those patients who do experience symptomatic relief following conventional anti-depressant treatment, clinical improvement is not evident for 3-4 weeks. Thus, there is a clear need to develop novel and improved therapeutics for unipolar depression.

A previous study showed that the intravenous administration of scopolamine produces antidepressant effects. This study is designed to determine if scopolamine combine with Escitalopram produce antidepressant effects at an early stage.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled clinical trial. Sixty-six outpatients (ages 18-45) with severe major depressive disorder (MDD) (17-item Hamilton Rating Scale for Depression total score greater than or equal to 20) are enrolled from Beijing Anding Hospital. All participants receive oral escitalopram 10 mg/d throughout the total of 4 weeks treatment. Meanwhile, they are randomized equally to one of three add-on treatment arms during the first three days: (1) intramuscular injection (i.m.) with saline (1 ml) at 9 am and 3 pm per day; (2) scopolamine (0.3 mg in 1ml saline, i.m.) at 9 am and saline (1 ml, i.m.) at 3 pm per day; (3) scopolamine (0.3 mg in 1ml saline, i.m.) at 9 am and 3 pm per day, respectively. Patients were assessed at baseline, day 2, day 3, day 4, day 7, day 14, and day 28 using 17-Item Hamilton Depression Rating Scale(HAMD-17), Montgomery-Asberg Depression Rating Scale(MADRS), Young Mania Rating Scale(YMRS), Generalized Anxiety Disorder-7(GAD-7), Quick Inventory of Depressive Symptomatology Self-report 16(QIDS-SR16) and Clinical Global Impression(CGI) by assessors masked to treatment assignments. The primary outcome measure was the time from randomization (baseline) to early improvement (at least 20% reduction in HAMD-17 score ). The second outcome measures were response rates (at least 50% decrease in the HAMD-17 at any visit from baseline), remission rate (HAMD-17 score≤7) at day 28, change in HAMD-17 score ,MADRS score, QIDS-SR16 score, GAD7 score and YMRS score from baseline to any visit, change in CGI-S from baseline to the end of the trial, and CGI-I score at any visit.

ELIGIBILITY:
Inclusion Criteria:

1. Has given written informed consent.
2. Male or female outpatients aged at least 18 years and not more than 45 years.
3. Has a diagnosis of major depressive disorder by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria.
4. Current HAMD-17 score ≥ 20 and the duration of the index episode is greater than or equal to four weeks.

Exclusion Criteria:

1. Currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an off-label use of an investigational drug.
2. Current Axis I primary psychiatric diagnosis other than major depressive disorder.
3. Organic mental disease, including mental retardation.
4. History of clinically significant disease, including any cardiovascular, hepatic, renal, respiratory, hematologic, endocrinologic, or neurologic disease, or clinically significant laboratory abnormality that is not stabilized or is anticipated to require treatment during the study.
5. Subjects receiving an investigational agent (including different formulation and generic agents of investigational drug) in the previous 3 months prior to screening.
6. Women in pregnancy or lactation, or female of child bearing potential without appropriate birth control measures.
7. Use of antipsychotics or mood stabilizers within 5 days prior to screening.
8. Has received depot antipsychotic medication within one cycle prior to screening.
9. Known allergy or lack of response to mirtazapine.
10. Has received ECT or MECT within 3 months prior to screening.
11. History of anticholinergic drug allergy or complications (allergic reaction, skin rash, urticaria and other allergic reactions which caused by drugs).
12. Smokers.
13. Significant risk of suicidal and/or self-harm behaviors

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
The time of early onset | From randomization (base line) to endpoint(Week 4)
  The time from randomization (baseline) to early improvement (at least 20% reduction in HAMD-17 score )

SECONDARY OUTCOMES:
Response rate of patients receiving scopolamine | From randomization (base line) to endpoint(Week 4)
  The proportion of subjects with at least 50% decrease in the HAMD-17 at any visit from baseline.Response was defined as ≥50% decrease in the baseline HAMD-17 total scores.
The proportion of subjects at endpoint with HAMD-17≤7 | endpoint(Week 4)
  Remission was defined as the HAMD total score ≤7
Change in 17-item Hamilton Depression Scale (HAMD-17) scores | From randomization (base line) to endpoint(Week 4)
  Change in HAMD-17 scores measured by the difference between baseline HAMD-17 score and HAMD-17 score at endpoint.
Change in Montgomery-Asberg Depression Rating Scale(MADRS) | From randomization (base line) to endpoint(Week 4)
  Change in MADRS scores measured by the difference between baseline MADRS score and MADRS score at endpoint.
Change in QIDS-SR16 score | From randomization (base line) to endpoint(Week 4)
  Change in QIDS-SR16 score measured by the difference between baseline QIDS-SR16 score and QIDS-SR16 score at endpoint.
Change in GAD7 score | From randomization (base line) to endpoint(Week 4)
  Change in GAD7 score measured by the difference between baseline GAD7 score and GAD7 score at endpoint.
Change in YMRS score | From randomization (base line) to endpoint(Week 4)
  Change in YMRS score measured by the difference between baseline YMRS score and YMRS score at endpoint.
Change in CGI-S score | From randomization (base line) to endpoint(Week 4)
  Change in CGI-S score measured by the difference between baseline CGI-S score and CGI-S score at endpoint.

OTHER OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability) | From randomization (base line) to endpoint(Week 4)
  The incidence and nature of overall adverse events; the incidence and nature of drug-related adverse events; assessment of cognitive function change by PDQ-D5

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, M.D.,Ph.D., Principal Investigator — Beijing Anding Hospital, Capital Medical University
Locations (1):
- Beijing Anding Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Furey ML, Drevets WC. Antidepressant efficacy of the antimuscarinic drug scopolamine: a randomized, placebo-controlled clinical trial. Arch Gen Psychiatry. 2006 Oct;63(10):1121-9. doi: 10.1001/archpsyc.63.10.1121. PMID 17015814
- [Derived] Zhou J, Yang J, Zhu X, Zghoul T, Feng L, Chen R, Wang G. The effects of intramuscular administration of scopolamine augmentation in moderate to severe major depressive disorder: a randomized, double-blind, placebo-controlled trial. Ther Adv Psychopharmacol. 2020 Jul 1;10:2045125320938556. doi: 10.1177/2045125320938556. eCollection 2020. PMID 32655854
- [Derived] Zhou J, Wang W, Yang J, Zhu X, Feng L, Xiao L, Wang G. Scopolamine augmentation of a newly initiated escitalopram treatment for major depressive disorder: study protocol for a randomized controlled trial. Trials. 2019 Jan 9;20(1):33. doi: 10.1186/s13063-018-3132-3. PMID 30626409
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/17015814